CLINICAL TRIAL: NCT02742441
Title: A Multicenter, Randomized, Double-Blind, Parallel Group Comparison of 122-0551 Foam Versus Vehicle Foam in Subjects With Plaque Psoriasis (Study 310)
Brief Title: A Comparison of 122-0551 Foam Versus Vehicle Foam in Subjects With Plaque Psoriasis (Study 310)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 122-0551-310
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 122-0551 Foam (Experimental): 122-0511 Foam, topically applied twice daily
  Intervention: Drug: 122-0551 Foam
  Interventions: Drug: 122-0551 Foam
- Vehicle Foam (Placebo Comparator): Vehicle Foam, topically applied twice daily
  Intervention: Drug: Vehicle Foam
  Interventions: Drug: Vehicle Foam

INTERVENTIONS:
Drug: 122-0551 Foam — Topical Foam containing active drug
  Arms: 122-0551 Foam
Drug: Vehicle Foam — Topical Foam containing no active drug
  Arms: Vehicle Foam

SUMMARY:
This Phase 3 study (Study 310) has been designed to determine and compare the efficacy and safety of 122-0551 Foam and Vehicle Foam applied twice daily for two weeks in subjects with plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or non-pregnant female and is at least 18 years of age at the time of the Screening Visit.
2. Subject has provided written informed consent.
3. Subject is willing and able to apply the test article(s) as directed, comply with study instructions and commit to all follow-up visits for the duration of the study.
4. Subject has a clinical diagnosis of stable plaque psoriasis involving a minimum of 2% and no more than 12% body surface area (BSA) (excluding the face, scalp, groin, axillae and other intertriginous areas).
5. Subject has an Investigator's Global Assessment (IGA) score of at least three (3 = moderate) at the Baseline Visit.
6. Females must be post-menopausal , surgically sterile or use an effective method of birth control , with a negative urine pregnancy test (UPT) at the Baseline Visit.

Exclusion Criteria:

1. Subject has spontaneously improving or rapidly deteriorating plaque psoriasis.
2. Subject has guttate, pustular, erythrodermic or other non-plaque forms of psoriasis.
3. Subject has a physical condition which, in the investigator's opinion, might impair evaluation of plaque psoriasis, or which exposes the subject to an unacceptable risk by study participation.
4. Subject has used any phototherapy (including laser), photo-chemotherapy or other forms of photo based therapy for the treatment of their psoriasis within 30 days prior to the Baseline Visit.
5. Subject has used any systemic methotrexate, retinoids, systemic corticosteroids [including intralesional, intra-articular, and intramuscular corticosteroids], cyclosporine or analogous products within 90 days prior to the Baseline Visit.
6. Subject has used any systemic biologic therapy (i.e., FDA-approved or experimental therapy) within five (5) half-lives of the biologic prior to the Baseline Visit. Published or documented half-life of the product provided by the commercial supplier or Sponsor should be used to establish this value.
7. Subject had prolonged exposure to natural or artificial sources of ultraviolet radiation within 30 days prior to the Baseline Visit or is intending to have such exposure during the study which in the opinion of the investigator is thought to modify the subject's disease.
8. Subject has used topical body (excluding the scalp) psoriasis therapy (including coal tar, anthralin, steroids, retinoids and vitamin D analogs) within 14 days prior to the Baseline Visit.
9. Subject has used emollients/moisturizers on areas to be treated within four hours prior to clinical evaluation at the Baseline Visit.
10. Subject is currently using lithium or Plaquenil (hydroxychloroquine).
11. Subject is currently using a beta-blocking medication (e.g., propranolol) or angiotensin converting enzyme (ACE) inhibitor at a dose that has not been stabilized, in the opinion of the investigator.
12. Subject has a history of sensitivity to any of the ingredients in the test articles.
13. Subject is pregnant, lactating, or is planning to become pregnant during the study.
14. Subject is currently enrolled in an investigational drug or device study.
15. Subject has used an investigational drug or investigational device treatment within 30 days prior to the Baseline Visit.
16. Subject has been previously enrolled in this study and treated with a test article.
17. Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol (e.g., due to alcoholism, drug dependency, mental incapacity) in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2016-06; Primary Completion 2017-02-27 (Actual); Study Completion 2017-06-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Site 14, Fort Smith, Arkansas
  - Site 01, Hot Springs, Arkansas
  - Site 17, Encino, California
  - Site 19, Denver, Colorado
  - Site 16, Brandon, Florida
  - Site 15, Clearwater, Florida
  - Site 20, Miami Lakes, Florida
  - Site 11, North Miami Beach, Florida
  - Site 12, Pinellas Park, Florida
  - Site 10, Carmel, Indiana
  - Site 06, New Albany, Indiana
  - Site 13, Quincy, Massachusetts
  - Site 07, Ann Arbor, Michigan
  - Site 02, Saint Joseph, Missouri
  - Site 08, Wilmington, North Carolina
  - Site 04, Gahanna, Ohio
  - Site 05, Nashville, Tennessee
  - Site 09, Austin, Texas
  - Site 18, San Antonio, Texas
  - Site 21, Norfolk, Virginia
  - Site 03, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bhatia N, Stein Gold L, Kircik LH, Schreiber R. Two Multicenter, Randomized, Double-Blind, Parallel Group Comparison Studies of a Novel Foam Formulation of Halobetasol Propionate, 0.05% vs Its Vehicle in Adult Subjects With Plaque Psoriasis. J Drugs Dermatol. 2019 Aug 1;18(8):790-796. PMID 31424709

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: June 2016 to February 2017
  The location of clinical sites included dermatology clinics and clinical research centers.
Pre-assignment Details: All subjects who met the entry criteria were randomized and enrolled into the study.
Groups:
- 122-0551 Foam: 122-0511 Foam, topically applied twice daily
  Intervention: Drug: 122-0551 Foam
  122-0551 Foam: Topical Foam containing active drug
- Vehicle Foam: Vehicle Foam, topically applied twice daily
  Intervention: Drug: Vehicle Foam
  Vehicle Foam: Topical Foam containing no active drug
Period: Overall Study
Arm/Group | 122-0551 Foam | Vehicle Foam
Started | 205 | 204
Completed | 199 | 196
Not Completed | 6 | 8
Not completed — Lost to Follow-up | 4 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 122-0551 Foam | Vehicle Foam | Total
Number analyzed (Participants) | 205 | 204 | 409
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (13.9) | 50.1 (14.0) | 50.2 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 86 | 178
  Male | 113 | 118 | 231
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 54 | 108
  Not Hispanic or Latino | 151 | 150 | 301
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 11 | 15 | 26
  White | 190 | 185 | 375
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 205 | 204 | 409

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Rated a "Treatment Success" Based on the Investigator's Global Assessment (IGA)
Description: The IGA score is a static evaluation of the overall or "average" degree of severity taking into account all of the subject's psoriatic lesions in the Treatment Area by the investigator or designee. This evaluation takes into consideration the three individual characteristics of psoriasis (scaling, erythema and plaque elevation) with the IGA score at each visit representing the average of scaling, erythema or plaque elevation that is present amongst all of the lesions eligible for treatment. IGA will be assessed on a 5-point scale where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe.
Time Frame: Day 15
Population: Analysis shown is based on the intent-to-treat population, defined as all enrolled participants who were randomized and applied at least one dose of the test article.
Measure: Number; unit: percentage of participants
Arm/Group | 122-0551 Foam | Vehicle Foam
Number analyzed (Participants) | 205 | 204
percentage of participants | 30.7 | 7.4
Statistical Analysis 1: Comparison: 122-0551 Foam vs Vehicle Foam; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Treatment groups were compared with respect to the proportions of subjects with "treatment success" at Day 15 using the Cochran-Mantel-Haenszel (CMH) test stratified by analysis center; Missing data was imputed as treatment failure

2. Secondary Outcome: Percentage of Subjects Rated a "Treatment Success" for Each of the Clinical Signs of Psoriasis (Scaling, Erythema and Plaque Elevation)
Description: Scaling, erythema and plaque elevation will each be scored on a 5-point scale where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe. These evaluations are an assessment of the overall or "average" degree of each of three key characteristics present within all of the subject's psoriatic lesions in the Treatment Area by the investigator or designee.
Time Frame: Day 15
Population: Analysis shown is based on the Intent-to-Treat (ITT) population.
Measure: Number; unit: percentage of participants
Arm/Group | 122-0551 Foam | Vehicle Foam
Number analyzed (Participants) | 205 | 204
percentage of participants
  Plaque Elevation | 35.0 | 9.9
  Scaling | 33.7 | 9.8
  Erythema | 28.8 | 8.3
Statistical Analysis 1: Comparison: 122-0551 Foam vs Vehicle Foam; Treatment groups were compared with respect to each of the clinical signs of psoriasis (plaque elevation, scaling, and erythema); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was achieved for each of the clinical signs of psoriasis; Missing data was imputed as treatment failure

3. Other Pre Specified Outcome: Percentage of Subjects Rated a "Treatment Success" Based on the Investigator's Global Assessment (IGA)
Time Frame: Day 8
Population: Analysis shown is based on the ITT population. Only participants with observed values are reported.
Measure: Number; unit: percentage of participants
Arm/Group | 122-0551 Foam | Vehicle Foam
Number analyzed (Participants) | 199 | 196
percentage of participants | 9.5 | 3.6
Statistical Analysis 1: Comparison: 122-0551 Foam vs Vehicle Foam; Test type: Superiority; p = 0.012, Cochran-Mantel-Haenszel

4. Other Pre Specified Outcome: Percentage of Subjects Rated a "Treatment Success" for Each of the Clinical Signs of Psoriasis (Scaling, Erythema and Plaque Elevation)
Time Frame: Day 8
Population: Analysis shown is based on the ITT population. Only participants with observed values are reported.
Measure: Number; unit: percentage of participants
Arm/Group | 122-0551 Foam | Vehicle Foam
Number analyzed (Participants) | 205 | 204
percentage of participants
  Plaque Elevation | 13.2 | 3.6
  Scaling | 14.2 | 3.6
  Erythema | 8.0 | 3.1

5. Other Pre Specified Outcome: Change From Baseline in Pruritus Score
Description: At the Baseline Visit, prior to the first application of the test article, the subject's overall experience of pruritus within the previous two (2) weeks will be assessed and scored (range 1-5) using a questionnaire that assesses the degree, duration, direction, disability, and distribution of the subject's pruritus. Possible total scores range from 5 (no pruritus) to 25 (most severe pruritus). At Day 15, the overall experience of pruritus, in the previous two weeks, will be scored using the same questionnaire.
Time Frame: Day 15
Population: Analysis shown is based on the ITT population. Only participants with observed values are reported. Pruritus scores were based on the patient's assessment of pruritus ranging from a score of 5 (no pruritus) to 25 (most severe pruritus).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | 122-0551 Foam | Vehicle Foam
Number analyzed (Participants) | 205 | 204
scores on a scale | -4.3 (3.8) | -2.5 (3.3)

6. Other Pre Specified Outcome: Changes in Percent BSA With Active Psoriasis in the Treatment Area
Description: The percent (%) Body Surface Area (BSA) with active psoriasis in the Treatment Area will be determined at the Baseline Visit and Week 2 (Day 15) and documented. At Baseline, the percent BSA with active psoriasis in the Treatment Area must be 2% to 12%, inclusive.
Time Frame: Day 15
Population: Analysis shown is based on the ITT population. Only participants with observed values are reported. The mean percent BSA with active psoriasis at Baseline was 5.4% and 5.1% for the active and vehicle groups, respectively.
Measure: Mean (Standard Deviation); unit: Change in percent BSA
Arm/Group | 122-0551 Foam | Vehicle Foam
Number analyzed (Participants) | 199 | 196
Change in percent BSA | -1.5 (2.3) | -0.2 (1.5)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from Study Day 1 (enrollment/first dose) to study completion (Day 15) or participant termination. AEs that continued beyond completion/termination were followed until resolution or stabilization.
Description: The safety population included all subjects enrolled in the study who were dispensed and applied the test article at least once; because the first dose of the test article was applied at the study site (Day 1), all enrolled subjects (N=409) were included in the safety population. Subjects reporting a particular AE more than once are counted only once for that AE.
Arm/Group | 122-0551 Foam | Vehicle Foam
All-Cause Mortality (participants affected / at risk) | 0/205 | 0/204
Serious Adverse Events (participants affected / at risk) | 0/205 | 1/204
Other Adverse Events (participants affected / at risk) | 12/205 | 14/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 122-0551 Foam (N=205) | Vehicle Foam (N=204)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) — The SAE was deemed unrelated to test article.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 122-0551 Foam (N=205) | Vehicle Foam (N=204)
Application site pain (General disorders) | 2 (2) | 1 (1)
Application site pruritis (General disorders) | 0 (0) | 2 (2)
Blepharitis (Eye disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has first right to publish pooled study data. In the event that such manuscript has not been submitted for publication within 12 months from study completion/termination at all participating sites, the PI shall have the right to single center publications provided they submit any data for presentation, oral or written, to the Sponsor for review 30 days prior to public disclosure. The PI may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT02742441/Prot_SAP_000.pdf